CLINICAL TRIAL: NCT04891549
Title: TENSION BAND VERSUS LOCKING PLATE FIXATION FOR THE TREATMENT OF PATELLA FRACTURE - a High Quality, Multicenter, Randomized Clinical Trial
Brief Title: Tension Band Versus Locking Plate Fixation for the Treatment of Patella Fractures
Acronym: TENPLA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rasmus Elsøe (Other)
Collaborators: Aarhus University Hospital (Other); Randers Regional Hospital (Other); Regional Hospital Hjoerring (Unknown); Regional Hospital Kolding (Unknown); Viborg Regional Hospital (Other)
Responsible Party: Sponsor-Investigator, Rasmus Elsøe, Head of orthopaedic trauma surgery, Aalborg University Hospital
Organization: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LERG2
Record Dates: First submitted 2021-05-13; First posted 2021-05-18 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Patella Fracture; Surgery; Orthopedic Disorder
Keywords: patella fracture; surgery; Tension band; Plate
MeSH Terms: conditions — Patella Fracture; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: This study is a multicenter pragmatic, prospective, assessor-blinded, randomized independent clinical trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Due to the surgical nature of the study the surgeon can not be blinded. The outcome assessor, patients and care providers will be blinded with regards to the two treatment groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tension band fixation (Active Comparator): Surgical fixation of the patella fracture utilizing the AO principles using K-wires, screws, cerclage and sutures by surgeons choice.
  Interventions: Procedure: Tension band fixation
- Plate fixation (Experimental): Surgical fixation of the patella fracture utilizing the AO principles and a locking plate with the number of screws by surgeons choice. Additional fixation by surgeons choice.
  Interventions: Procedure: Plate fixation

INTERVENTIONS:
Procedure: Tension band fixation — Fracture fixation of the patella fracture with tension band.
  Arms: Tension band fixation
Procedure: Plate fixation — Fracture fixation of the patella fracture with a plate.
  Arms: Plate fixation

SUMMARY:
This study is a multicenter pragmatic, prospective, assessor-blinded, randomized independent clinical trial in which we compare locking plate fixation to standard tension band fixation in patients with patella fractures.

DETAILED DESCRIPTION:
This study is a multicenter pragmatic, prospective, assessor-blinded, randomized independent clinical trial in which we compare locking plate fixation to standard tension band fixation in patients with patella fractures.

Primary objective The overall objective of the study is to compare the 1-year patient-reported Knee Injury and Osteoarthritis Outcome Score (KOOS5) after standard tension band fixation with locking plat fixation for patients with patella fractures.

Secondary objectives Several other analyses are of interest and are planned but are not objectives of this study. Therefore, these analyses will, for the major part, hypothesis-generating. Analyses of this type include, but are not limited to harms, muscle atrophy, pain, general health, gait function, time to return to work and economical consequences between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years of age
* Patella fracture suitable for surgically treatment, with both surgical methods
* AO classification 34-B, 34-C

Exclusion Criteria:

* Open patella fracture above Gustillo grade 2
* Bilateral patella fracture
* Total knee replacement in the affected extremity
* Other fractures of the affected extremity within the previous 12 months.
* Other reasons for exclusion (unable to understand Danish, mentally unable to participate, etc).
* Prior ipsilateral patella fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score - (KOOS5) | One year following treatment
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) 29 is a standardised patient-reported questionnaire developed to evaluate knee problems. The questionnaire includes five subscales: pain, ADL, symptoms, sport and QOL and an overall score KOOS 5 subscales.

SECONDARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score - (KOOS5) | 3- and 6 months
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) 29 is a standardised patient-reported questionnaire developed to evaluate knee problems. The questionnaire includes five subscales: pain, ADL, symptoms, sport and QOL and an overall score KOOS5 can be calculated. A total score of 100 indicates no symptoms, and 0 indicates major symptoms.
Knee Injury and Osteoarthritis Outcome Score - subscales: pain, ADL, symptoms, sport and QOL. | 3-, 6- and 12-months
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) 29 is a standardised patient-reported questionnaire developed to evaluate knee problems. The questionnaire includes five subscales: pain, ADL, symptoms, sport and QOL and an overall score KOOS5 can be calculated. A total score of 100 indicates no symptoms, and 0 indicates major symptoms.
EQ-5D-5L questionnaire (5-level version) | 3-, 6- and 12-months
  General health will be assessed using EQ-5D-5L questionnaire (5-level version), both the descriptive index and the EQ-VAS. It consists of five dimensions: Mobility, self-care, usual activities, pain/discomfort and anxiety/depression, and a self-rated health scale on a 20 cm vertical, visual analogue scale with endpoints labelled 'the best health you can imagine' and 'the worst health you can imagine'. An Eq5d-5L index of 1.0 indicated full health, 0 death, and -0.59 denoted a condition worse than death.
Pain intensity measured on a 10 cm VAS scale | 3-, 6- and 12-months
  Development in pain will be recorded by patient-reported pain intensity measured on a 10 cm visual analogue scale (VAS) with endpoints "no pain" and "maximal pain" for the worst pain during the last 24 hours and resting pain.
"PainDETECT" questionnaire | 3-, 6- and 12-months
  Knee pain and neuropathic pain will be assessed using the "PainDETECT" questionnaire. The "PainDETECT" screening questionnaire uses a scoring method between 1-38. A total score of 1 indicates no symptoms, and 38 indicates major symptoms.
Bone union | 3-, 6- and 12-months
  Bone union, will be evaluated on standard AP and side X-rays of the fractured patella. The evaluation of bone union will be defined as: i) visible callus formation, diminished no visible fracture line and no pain from the fracture site at weight-bearing and at clinical examination.
Maximum isometric knee-extension strength | 12-months
  Maximum isometric knee-extension strength at 60 degrees knee flexion measured as Nm/kg body mass. Will be measured bilaterally by a strap-mounted dynamometer attached to the wall (Mecmesin AFG2500, Mecmesin Ltd, West Sussex, UK)
Maximum isometric knee-flexion strength | 12-months
  Maximum isometric knee-flexion strength at 90 degrees knee flexion measured as Nm/kg body mass. Will be measured bilaterally by a strap-mounted dynamometer attached to the wall (Mecmesin AFG2500, Mecmesin Ltd, West Sussex, UK)
Knee range of motion | 3-, 6- and 12-months
  Knee range of motion. With the patient supine on an examination table the full range of passive motion in both knee joints will be measured using a standard goniometer.
Time to return to work | 3-, 6- and 12-months
  Measure the time from surgery to end of sick leave measured in days

OTHER OUTCOMES:
Harms | 3-, 6- and 12-months
  Adverse events, defined as any negative or unwanted reactions to the two groups will be recorded. Based on previous reports we will focus on: infection, DVT and re-operation. Patients are continuously requested to report any suspicion of a potential AE. Furthermore, adverse events (AE) will be recorded at 3-, 6- and 12-months follow-up by asking patients about potential AEs using open-probe questioning to ensure that all AEs are recorded. Furthermore, medical records will be checked at the primary endpoint (12 months) for all AEs occurring from inclusion until the 12 months follow-up. An AE is defined as any undesirable experience during follow-up leading to contact with the healthcare system (general practitioner or hospital). If an AE result in hospitalization, prolonged inpatient hospital care, result in re-surgery, or if an AE is life-threatening, result in death, permanent disability or damage, they will be categorized as serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Rasmus Elsoe, MD, PhD, Study Chair — Aalborg University Hospital, Denmark; Peter Larsen, PT, PhD, Principal Investigator — Aalborg University Hospital, Denmark
Locations (6):
- Denmark (6):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Regional Hospital Hjoerring, Hjørring
  - Regional Hospital Kolding, Kolding
  - Regional Hospital Randers, Randers
  - Regional Hospital Viborg, Viborg

IPD SHARING:
Plan to Share IPD: No
A detailed statistical analysis plan will be made publicly available before the last patient is included in the study.

REFERENCES:
- [Derived] Elsoe R, Thorninger R, Severinsen R, Beuke JC, Serritslev R, Jensen SS, Rasmussen MK, Szephalmi P, Petruskevicius J, Barckman J, Bruun NH, Larsen P. Tension band versus locking plate fixation for patella fractures - a protocol of a randomised controlled trial. Dan Med J. 2024 Apr 10;71(5):A12230753. doi: 10.61409/A12230753. PMID 38704836
- See also: The full study protocol are published online before study start — https://vbn.aau.dk/ws/portalfiles/portal/410910476/Protokol_patella_multicenter_final_version_16042021.pdf